CLINICAL TRIAL: NCT02784080
Title: Donor Specific HLA Alloantibodies in Liver Transplantation: a Prospective Blinded Multicenter Prognostic Study
Brief Title: Donor Specific HLA Alloantibodies in Liver Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Sahlgrenska University Hospital (Other); Karolinska Institutet (Other); Helsinki University Central Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Arendtsen Rostved, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: H-15007823
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Complication of Transplanted Liver
Keywords: Liver Transplantation; HLA alloantibodies; donor specific antibodies; Mortality; Re-transplantation; Rejection; Acute rejection; Chronic rejection; Biliary complications; Biliary stricture; Arterial thrombosis; Arterial stenosis; Portal vein thrombosis; Fibrosis; Single antigen bead; Cross-match
MeSH Terms: conditions — Rejection, Psychology; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Recipient samples, pre-transplant, at discharge or day 14 (±4 days, changed to discharge), 3 months (±3 weeks), 1 year (±1 month), and at liver biopsy
  * 1 Plasma, EDTA-glass (9 ml), redistributed 4 aliquots
  * 2 Serum, clot activator (9 ml + 4 ml), redistributed 8 aliquots
  * Liver biopsy sample: Formalin fixed paraffin-embeded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HLA-alloantibodies exposure: Preformed, persistent, and de novo HLA-alloantibody exposure in the whole cohort.
  Interventions: Other: HLA-alloantibodies exposure

INTERVENTIONS:
Other: HLA-alloantibodies exposure — Following analyzes will be done:
  LABScreen® Single Antigen, One Lambda, CA
  C1qScren™, One Lambda, CA (planned for later study)
  PE-conjugated IgG3 antibody (planned for later study)
  LABScreen® Mixed, One Lambda, CA (never analysed in the study)

SUMMARY:
The aim is to evaluate the impact of donor specific HLA alloantibodies (DSA) on all-cause mortality and re-transplantation, early allograft dysfunction, acute and chronic rejection, fibrosis, vascular, and biliary complications. Furthermore, all biopsies will be C4d stained. The hypothesizes is that donor specific HLA alloantibodies facilitate an immune mediated damage to the liver allograft that impairs function and lead to various complications.

The investigators will do a prospective blinded multicenter cohort study in the Scandiatransplant organ sharing organization region.

Both preformed, persistent, and de novo donor specific HLA alloantibodies will studied. Blood samples will be taken immediately prior to transplantation, and 14 days, 3 months, and 1 year after transplantation. All liver biopsies performed during the study period will be evaluated for a humoral component and blood samples will be obtained prior to liver biopsies to investigate the presence of DSA.

Investigations will be fully blinded for the treatment responsible doctors.

DETAILED DESCRIPTION:
The outcome after liver transplantation has improved drastically over time, but this development has stagnated in recent years to a graft failure rate of 9-15 % within the first year and approximately 20-30 % at 5 years [1]. The primary goal is to improve the outcome after liver transplantation.

The impact of donor specific antibodies (DSA) on all-cause mortality and re-transplantation, early allograft dysfunction, acute and chronic rejection, vascular and biliary complications and fibrosis will be investigated.

Objectives:

1. The primary objective is to investigate if DSA both pre-formed, persistent, and de novo affect survival and allograft loss. For patients diagnosed with HLA antibodies a standard Luminex single antigen IgG analysis, a Luminex C1q and an IgG3 single antigen assay will be performed.
2. The secondary objective is to investigate if donor specific antibodies, both pre-formed, persistent, and de novo increase the risk of early allograft dysfunction, acute and chronic rejection, fibrosis, de novo autoimmune hepatitis (pediatric patients only), vascular and biliary complications. All liver biopsies will be stained by C4d and a DSA analysis will be undertaken.
3. Continuous measurements will be used to establish the kinetics of both preformed og de novo DSA after liver transplantation.

Pediatric patients will be analyzed separately.

In 2021 it was decided to split the study in a preformed and de novo study.

Preformed DSA

1. Our primary objective is to investigate if preformed and persistent DSA class I and II affect survival and re-transplantation.
2. The secondary objective is to investigate if preformed and persistent DSA class I and II is correlated with increased risk of acute rejection and early allograft dysfunction.

Preformed DSA will be analysed in 4 different ways separately for donor specific HLA class I and class II antibodies.

1. Dichotomous analysis defined as any DSA class I or II MFI >1000 is considered positive.
2. Number of different class I or II DSA will be analyzed as an ordinal variable.
3. A continuous variable by MFI, as a sum of all. Homozygous donors will not be accounted for.
4. Analysis will be done for no antibodies versus: 1) HLA-DQ (including DRB5 subtypes) 2) HLA-DR 3) HLA-DQ and -DR. Both as categorical and binary.

ELIGIBILITY:
Inclusion Criteria:

* Undergo a liver transplanted during the study period.
* Pre-transplant serum sample of minimum 4 ml (relevant for pediatric patients)
* Informed consent is given.

Exclusion Criteria:

* Withdrawal of informed consent.
* Blinding broken in a non-protocoled manner the patient will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All liver transplant recipients, both children and adults, in the Scandiatransplant region. The Scandiatransplant is an organ exchange organization that comprise of five centers in the Nordic countries: Norway, Sweden, Finland and Denmark. The five centers cover the need for liver transplantation in approximately 25 million people. From 2010-2015 the following number of transplants were done in Scandiatransplant according to the number of available donors: 323, 352, 353, 365, 388, and 401.
  Preliminary sample size calculations have estimated inclusion of 1062 adult and 100 pediatric patients during a study period of 3 years. Interim sample size calculations will be done, if necessary the study period will be prolonged.
  Pediatric patients will be analyzed separately.
Sampling Method: Probability Sample
Enrollment: 858 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or re-transplantation (graft loss) | Minimum 1 year, accrual to study end

SECONDARY OUTCOMES:
Early allograft dysfunction are defined as total bilirubin >10 mg/dl or INR >1.6 at day 7 after liver transplantation or ALT >2000 IU/L within the first 7 days after liver transplantation. | 7 days after transplantation
Acute rejection, both cellular and humoral rejection, as defined by Banff classification. | Minimum 1 year, accrual to study end
Chronic rejection, as defined by Banff classification, and as proposed by O'leary et al "Proposed Diagnostic Criteria for Chronic Antibody-Mediated Rejection in Liver Allografts". | Minimum 1 year, accrual to study end
Fibrosis, defined by METAVIR score. | Minimum 1 year, accrual to study end
Vascular complications (hepatic arterial stenosis, hepatic arterial thrombosis, portal vein thrombosis). | Minimum 1 year, accrual to study end
Biliary complications (biliary leakage, anastomotic biliary stricture, non-anastomotic biliary stricture, liver abscess, cholangitis, other). | Minimum 1 year, accrual to study end
  Anastomotic strictures and non-anastomotic strictures will be investigated as a combined and solitary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Rasmussen, MD, Study Chair — Department of Surgical Gastroenterology and Transplantation, Rigshospitalet - Copenhagen University Hospital, Denmark; Andreas A Rostved, MD, Principal Investigator — Department of Surgical Gastroenterology and Transplantation, Rigshospitalet - Copenhagen University Hospital, Denmark; Helle Bruunsgaard, MD, DMSc, Study Director — Department of Clinical Immunology, Centre of Diagnostic Investigation, Rigshospitalet - Copenhagen University Hospital
Locations (5):
- Department of Surgical Gastroenterology and Transplantation, Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Transplantation and Liver Surgery Clinic, Helsinki University Hospital, Helsinki, Finland
- Department of Transplantation Medicine, Oslo University Hospital, Oslo, Norway
- Sweden (2):
  - Surgery Department, Transplantation and Liver Surgery Unit, Sahlgrenska University Hospital, Gothenburg
  - Division of Transplantation Surgery, Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim WR, Smith JM, Skeans MA, Schladt DP, Schnitzler MA, Edwards EB, Harper AM, Wainright JL, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2012 Annual Data Report: liver. Am J Transplant. 2014 Jan;14 Suppl 1:69-96. doi: 10.1111/ajt.12581. PMID 24373168